CLINICAL TRIAL: NCT04262206
Title: PRagmatic EValuation of evENTs And Benefits of Lipid-lowering in oldEr Adults (PREVENTABLE)
Brief Title: Pragmatic Evaluation of Events And Benefits of Lipid-lowering in Older Adults
Acronym: PREVENTABLE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pro00103844; 1U19AG065188-01 (NIH)
Record Dates: First submitted 2020-02-07; First posted 2020-02-10 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-06

CONDITIONS: Cognitive Impairment, Mild; Dementia; Cardiovascular Diseases
Keywords: statin; older adults
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Cardiovascular Diseases | interventions — Atorvastatin; Tablets

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 atorvastatin 40mg vs. placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- atorvastatin 40mg (Experimental): 40mg atorvastatin po qd from consent to study end
  Interventions: Drug: Atorvastatin 40 Mg Oral Tablet
- Placebo (Placebo Comparator): matching placebo po qd from consent to study end
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Atorvastatin 40 Mg Oral Tablet — To generate knowledge about the role of statins in older adults in whom risk/benefit for primary prevention is understudied,
  Other Names: Lipitor
  Arms: atorvastatin 40mg
Drug: Placebo oral tablet — To generate knowledge about the role of statins in older adults in whom risk/benefit for primary prevention is understudied,
  Arms: Placebo

SUMMARY:
PREVENTABLE is a multi-center, randomized, parallel group, placebo-controlled superiority study. Participants will be randomized 1:1 to atorvastatin 40 mg or placebo. This large study conducted in community-dwelling older adults without cardiovascular disease (CVD) or dementia will demonstrate the benefit of statins for reducing the primary composite of death, dementia, and persistent disability and secondary composites including mild cognitive impairment (MCI) and cardiovascular events.

DETAILED DESCRIPTION:
PREVENTABLE will randomly assign atorvastatin 40 mg daily or matching placebo daily to approximately 20,000 community-dwelling adults 75 years of age or older without clinically evident cardiovascular disease, significant disability, or dementia, and follow them for up to 5 years (estimated median of 3.8 years). The study will enroll participants from approximately 100 US sites. Community engagement efforts will leverage community groups and practices as collaborators for recruitment. We plan to partner with participants, caregivers, and clinicians in all aspects of the study. The enrolling sites are non-VA and VA sites. To assist in recruitment, sites will apply a study-specific cohort identification algorithm to their electronic health record to create a list of eligible participants based on study inclusion and exclusion criteria. The cohort identification will exclude individuals with clinically evident cardiovascular disease, significant disability, or dementia and other exclusions obtainable from data queries to define a potential cohort. Additionally, the PREVENTABLE CCC will provide a centralized support team to assist with recruitment and retention efforts. This includes mass mailings and/or phone calls to potential participants and a toll-free number for potential participants to call for information and pre-screening. Interested and potentially eligible participants will be referred to an enrolling site near them, if applicable, otherwise, they will be referred to the PREVENTABLE Telesite which is capable of enrolling English and Spanish-speaking participants across the U.S. remotely. Sites will screen potential participants to confirm eligibility and consent and randomize those interested in joining the study. Specifically related to dementia, the qualifying exclusion is a clinical diagnosis in the chart or clinician's assessment that dementia may be present.

Sites will enter contact information, mailing address for study drug, demographic information, height, weight, statin history (if any), Social Security Number, and aspects of the medical history not obtainable from EHR. In addition, a Short Physical Performance Battery (SPPB) and Activities of Daily Living (ADL) screen will be site-performed at baseline. SPPB will provide an objective assessment of function for understanding frailty and physical function of the enrolled population. Baseline lipid panel (core lab) and biospecimen samples will be obtained using the same blood draw for 20cc of blood. Blinded lipid testing will be performed at baseline on all participants (n=20,000) and repeated at 3 months in a random subset (n=2,000). Lipid panels will be sent to the PREVENTABLE Core Lab to maintain study blind. Future testing of lipid panels during routine clinical care will be actively discouraged, but other laboratory testing as indicated by clinical care is permitted. Sites will have the option for telehealth enrollment. Baseline SPPB and Biorepository Labs are not required, but encouraged.

As part of the study operations, with the rationale of providing patient centricity, ease of participation, and access for vulnerable and at risk participants, follow up will be performed by a central call center. The baseline and annual assessments performed centrally will include a phone screen for cognitive function (TICS-M) and physical function (Patient-reported Outcome Measurement Information System-Physical Function [PROMIS-PF]). After year 1, if baseline calls indicated by crossing pre-specified cutpoints, in-person assessments will be completed by trained and certified research staff at a mutually agreed upon time and a standardized interview of a knowledgeable informant. Cardiovascular event ascertainment will be via a systematic approach to data curation from the EHR, Medicare, and National Death Index. For convenience and compliance, the study pharmacy will mail a supply of study drug, sufficient for 90 days, directly to participants. This will start immediately after randomization and continue as long as the participant is on study drug.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults
* Age ≥75 years
* English or Spanish as primary language
* Able to provide a trusted contact

Exclusion Criteria:

* Clinically evident cardiovascular disease defined as prior myocardial Infarction (MI), prior stroke, prior revascularization procedure, or a secondary prevention indication for a statin (clinician determined)
* Hospitalization for a primary diagnosis of heart failure in the prior 12 months (Note: History of heart failure in the absence of recent hospitalization or clinically evident cardiovascular disease is not an exclusion)
* Dementia (clinically evident or previously diagnosed)
* Dependence in any Katz Basic Activities of Daily Living [ADL] (with the exception of urinary or bowel continence)
* Severe hearing impairment (preventing phone follow up)
* Unable to talk (preventing phone follow up)
* Statin use in the past year or for longer than 5 years previously (participant reported)
* Ineligible to take atorvastatin 40 mg (clinician determined)
* Documented intolerance to statins
* Active Liver Disease

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients without diagnosis of new dementia | 4 years
  Number of patients without diagnosis of new dementia in each group (placebo vs. atorvastatin)
Number of patients without of persistent disability | 4 years
  Number of patients without chronic disability in each group

SECONDARY OUTCOMES:
Cardiovascular mortality measured as a composite of CV death, hospitalization for myocardial infarction/unstable angina, heart failure, stroke/TIA, or coronary revascularization | 4 years
  Cardiovascular mortality is measured by a composite measure of multiple CV conditions.
Cognitive disability as measured as a composite of MCI or probable dementia | 4 years
  Cognitive disability is measured by a composite of having mild cognitive impairment or probable dementia.

CONTACTS AND LOCATIONS:
Locations (103):
- United States (102):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Birmingham VA, Birmingham, Alabama
  - Southern Arizona VA Health Care System - Tucson, Tucson, Arizona
  - Little Rock VA Medical Center, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Fresno VA Medical Center, Fresno, California
  - Long Beach VA Medical Center, Long Beach, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - VA Greater Los Angeles, Los Angeles, California
  - VA Palo Alto Healthcare System, Palo Alto, California
  - VA San Diego Medical Center, San Diego, California
  - Yale University, New Haven, Connecticut
  - VA Connecticut Healthcare System, West Haven, Connecticut
  - Bay Pines VA, Bay Pines, Florida
  - Gainesville VA Medical Center, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - University of Florida, Jacksonville, Florida
  - Miami VA Medical Center, Miami, Florida
  - University of Miami, Miami, Florida
  - Atlanta VA Medical Center, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Chicago VA Medical Center/Jesse Brown VA, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Hines VA Medical Center, Hines, Illinois
  - North Chicago VA Medical Center, North Chicago, Illinois
  - Indianapolis VA Medical Center, Indianapolis, Indiana
  - University of Iowa Healthcare, Iowa City, Iowa
  - Kansas City VA Medical Center, Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - VA Eastern Kansas Healthcare System, Topeka, Kansas
  - Louisville VA Medical Center, Louisville, Kentucky
  - University Medical Center, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Maine VA Health Care System, Togus, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - VA Boston Healthcare System, Boston, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Essentia Health, Duluth, Minnesota
  - Allina Health, Minneapolis, Minnesota
  - Minneapolis VA Health Care System, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - VA Medical Center Jackson, Jackson, Mississippi
  - University of Missouri Health System, Columbia, Missouri
  - St. Louis VA Medical Center, St Louis, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Omaha VA Medical Center, Omaha, Nebraska
  - Reno VA/Sierra Nevada Health Care, Reno, Nevada
  - Northwell Health, Manhasset, New York
  - VA Hudson Valley Healthcare System, Montrose, New York
  - VA New York Harbor Healthcare System, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Bronx VA Medical Center, The Bronx, New York
  - Asheville VA-Charles George VA Medical Center, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Atrium Health, Charlotte, North Carolina
  - PREVENTABLE Tele-Site, Durham, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Duke University - Kannapolis, Kannapolis, North Carolina
  - Wake Forest Baptist Hospital-Cardiology, Winston-Salem, North Carolina
  - Wake Forest Hospital - Geriatrics, Winston-Salem, North Carolina
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Dayton VA Medical Center, Dayton, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Corporal Michael J. Crescenz VA Medical Center-Philadelphia VA, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Providence VA Medical Center, Providence, Rhode Island
  - Charleston VA Medical Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Columbia VA Health Care/Dorn VA Medical Center, Columbia, South Carolina
  - VA Medical Center Memphis, Memphis, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Nashville VA Medical Center, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Scott and White Medical Center, Dallas, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center Dallas, Dallas, Texas
  - Doctors Hospital at Renaissance, Edinburg, Texas
  - University of Texas at Houston, Houston, Texas
  - San Antonio VA Medical Center, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Intermountain, Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - VA Salt Lake City Healthcare System, Salt Lake City, Utah
  - Richmond VA, Richmond, Virginia
  - Clarksburg VA Medical Center, Clarksburg, West Virginia
  - Mayo Clinic Health Systems - NW Wisconsin, Eau Claire, Wisconsin
  - Mayo Clinic Health System SW Wisconsin, La Crosse, Wisconsin
  - VA Madison Healthcare System, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Milwaukee VA Medical Center, Milwaukee, Wisconsin
- VA Carribbean Healthcare, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Speiser JL, Ambrosius WT, Pajewski NM. Performance of Cox regression models for composite time-to-event endpoints with component-wise censoring in randomized trials. Clin Trials. 2023 Oct;20(5):507-516. doi: 10.1177/17407745231177046. Epub 2023 May 26. PMID 37243355
- [Derived] Joseph J, Pajewski NM, Dolor RJ, Sellers MA, Perdue LH, Peeples SR, Henrie AM, Woolard N, Jones WS, Benziger CP, Orkaby AR, Mixon AS, VanWormer JJ, Shapiro MD, Kistler CE, Polonsky TS, Chatterjee R, Chamberlain AM, Forman DE, Knowlton KU, Gill TM, Newby LK, Hammill BG, Cicek MS, Williams NA, Decker JE, Ou J, Rubinstein J, Choudhary G, Gazmuri RJ, Schmader KE, Roumie CL, Vaughan CP, Effron MB, Cooper-DeHoff RM, Supiano MA, Shah RC, Whittle JC, Hernandez AF, Ambrosius WT, Williamson JD, Alexander KP; PREVENTABLE Trial Research Group. Pragmatic evaluation of events and benefits of lipid lowering in older adults (PREVENTABLE): Trial design and rationale. J Am Geriatr Soc. 2023 Jun;71(6):1701-1713. doi: 10.1111/jgs.18312. Epub 2023 Apr 20. PMID 37082807
- [Derived] Rozing MP, Westendorp RGJ. Altered cardiovascular risk pattern of LDL cholesterol in older adults. Curr Opin Lipidol. 2023 Feb 1;34(1):22-26. doi: 10.1097/MOL.0000000000000859. Epub 2022 Nov 16. PMID 36413436